CLINICAL TRIAL: NCT07287761
Title: Comparison of Erector Spinae Plane Block and Serratus Posterior Superior Intercostal Plane Block in Postoperative Pain Management After Coronary Artery Bypass Grafting: A Prospective, Observational Study
Brief Title: Comparison of Erector Spinae Plane Block and Serratus Posterior Superior Intercostal Plane Block in Postoperative Pain Management After Coronary Artery Bypass Grafting
Status: Recruiting | Type: Observational
Sponsor: Ankara Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Abdullah KONAN, Principal Investigator, Ankara Education and Research Hospital
Other Study IDs: 496
Record Dates: First submitted 2025-11-25; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Pain After Thoracic Surgery; Coronary Artery Bypass Graft (CABG)
Keywords: Erector Spinae Plane Block (ESPB); Regional Anesthesia; Post-CABG Pain; Postoperative pain; Coronary Artery Bypass Graft Surgery; Serratus Posterior Superior Intercostal Plane Block (SPSIPB)
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ESPB Group: Erector Spinae Plane Block (ESPB) with Bupivacaine
- SPSIPB Group: Serratus Posterior Superior Intercostal Plane Block (SPSIPB) with Bupivacaine

SUMMARY:
Coronary Artery Bypass Grafting (CABG) is a common surgical procedure for ischemic heart disease, but it often leads to severe acute and chronic postoperative pain, which can delay recovery and reduce patient comfort. Effective pain management is crucial to prevent pulmonary complications and long hospital stays. Peripheral nerve blocks are increasingly used to reduce opioid consumption and improve patient satisfaction after major surgery.

This prospective, observational study aims to compare the effectiveness and safety of two different regional anesthesia techniques, the Erector Spinae Plane Block (ESPB) and the Serratus Posterior Superior Intercostal Plane Block (SPSIPB), in managing postoperative pain in patients undergoing CABG via median sternotomy.

Patients aged 18-80 years, classified as ASA II-III, who are scheduled for elective CABG will be included. The choice of block technique (ESPB or SPSIPB) will be determined by the operating anesthesiologist based on the visibility of anatomical structures (transverse processes) under ultrasound guidance. All patients will receive the same general anesthesia and be managed postoperatively with Intravenous Patient-Controlled Analgesia (PCA).

The main goal is to determine which block provides optimal pain control, measured by the time to first rescue analgesia and pain scores (NRS) at various time points after extubation. Secondary outcomes include intraoperative opioid consumption, total PCA usage, extubation time, and the incidence of opioid-related side effects. The findings will help optimize pain protocols for cardiac surgery patients.

DETAILED DESCRIPTION:
This is a single-center, prospective, observational study conducted at the University of Health Sciences Ankara Training and Research Hospital. The primary clinical challenge addressed is the intense postoperative pain following median sternotomy for Coronary Artery Bypass Grafting (CABG), which requires multimodal analgesia. The use of ultrasound-guided interfascial plane blocks has gained popularity due to their ease of application and lower complication rates compared to traditional methods.

Rationale for Comparison:

The Erector Spinae Plane Block (ESPB) has proven efficacy in thoracic and abdominal procedures. The Serratus Posterior Superior Intercostal Plane Block (SPSIPB) is being investigated as a potential alternative, targeting a broader area to manage pain in cardiac surgery. The study aims to provide clinical evidence regarding which of these two specific regional techniques offers superior postoperative pain control in this patient population.

Procedure Detail (Specific to Observation):

The selection of the block type (ESPB or SPSIPB) for the patient is determined intraoperatively by the experienced anesthesiologist based on the quality of the ultrasound image (visibility of the transverse processes) to ensure the most anatomically suitable block is performed.

Anesthesia Protocol (Standardized):

All enrolled patients (ASA II-III) will receive the same general anesthesia protocol (Thiopental, Fentanyl, Rocuronium for induction; Sevoflurane for maintenance). The regional block will be administered by a single experienced anesthesiologist under the supervision of the responsible investigator, using a bilateral injection of 30 mL of 0.25% Bupivacaine for both techniques. Postoperative analgesia will be managed using a standardized Intravenous Patient-Controlled Analgesia (PCA) device, set at a 3mg/ml concentration, with a 24mg bolus dose and a 20-minute lockout interval.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective Coronary Artery Bypass Grafting (CABG) via median sternotomy.
* Age between 18 and 80 years.
* Classification of American Society of Anesthesiologists (ASA) Physical Status Class II or III.
* Patients who provide written and verbal informed consent to participate in the study.

Exclusion Criteria:

* Patients who do not provide consent.
* Age older than 80 years or ASA Physical Status Class > III.
* Patients who do not understand the Numerical Rating Scale (NRS) or have communication difficulties.
* Patients with a known history of coagulation disorders or bleeding disorders.
* Patients with skin infection at the site of peripheral nerve block application.
* Patients with Morbid Obesity (Body Mass Index BMI>35 kg/m2).
* Patients with chronic pain, opioid or substance dependence, or who use chronic analgesics.
* Patients with known allergy to local anesthetics.
* Patients with liver or kidney function disorders.
* Patients with a history of previous median sternotomy operation.
* Patients undergoing emergency surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients (18 to 80 years) classified as ASA Physical Status Class II or III, who are scheduled to undergo elective Coronary Artery Bypass Grafting (CABG) requiring median sternotomy at the University of Health Sciences Ankara Training and Research Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Total Opioid Consumption in the Perioperative Period | Up to 24 hours post-extubation
  The cumulative dose of all opioids administered (Intraoperative Fentanyl and Post-Extubation Tramadol via PCA and rescue doses of Morphine) will be calculated in Morphine Equivalent Dose (mg).

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Training and Research Hospital, Ankara, Altındag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the results reported in this article (such as anonymized patient-level data, study protocol, statistical analysis plan) will be shared. Data will be made available to researchers who provide a methodologically sound proposal for research and sign a data access agreement. Access will be provided after the article is published and for a period of 5 years following publication
Supporting Information: Study Protocol, SAP
Time Frame: Data will be made available beginning 6 months after publication of the main results in a peer-reviewed journal and will remain available for a period of 5 years after the publication date.
Access Criteria: Access will be granted to researchers who submit a methodologically sound proposal for research purposes. The requester must sign a Data Sharing Agreement guaranteeing the use of the data will be restricted to the proposed research and that the anonymity of participants will be protected. Data will be provided in an anonymized, de-identified format.

REFERENCES:
- [Background] Tulgar S, Ciftci B, Ahiskalioglu A, Bilal B, Sakul BU, Korkmaz AO, Bozkurt NN, De Cassai A, Torres AJ, Elsharkawy H, Alici HA. Serratus Posterior Superior Intercostal Plane Block: A Technical Report on the Description of a Novel Periparavertebral Block for Thoracic Pain. Cureus. 2023 Feb 3;15(2):e34582. doi: 10.7759/cureus.34582. eCollection 2023 Feb. PMID 36883093
- [Background] Rothaug J, Zaslansky R, Schwenkglenks M, Komann M, Allvin R, Backstrom R, Brill S, Buchholz I, Engel C, Fletcher D, Fodor L, Funk P, Gerbershagen HJ, Gordon DB, Konrad C, Kopf A, Leykin Y, Pogatzki-Zahn E, Puig M, Rawal N, Taylor RS, Ullrich K, Volk T, Yahiaoui-Doktor M, Meissner W. Patients' perception of postoperative pain management: validation of the International Pain Outcomes (IPO) questionnaire. J Pain. 2013 Nov;14(11):1361-70. doi: 10.1016/j.jpain.2013.05.016. Epub 2013 Sep 7. PMID 24021577
- [Background] Wang AH, Juan AH, Ko KD, Tsai PF, Zare H, Dell'Orso S, Sartorelli V. The Elongation Factor Spt6 Maintains ESC Pluripotency by Controlling Super-Enhancers and Counteracting Polycomb Proteins. Mol Cell. 2017 Oct 19;68(2):398-413.e6. doi: 10.1016/j.molcel.2017.09.016. Epub 2017 Oct 12. PMID 29033324
- [Background] Mazzeffi M, Khelemsky Y. Poststernotomy pain: a clinical review. J Cardiothorac Vasc Anesth. 2011 Dec;25(6):1163-78. doi: 10.1053/j.jvca.2011.08.001. Epub 2011 Sep 29. No abstract available. PMID 21955825